CLINICAL TRIAL: NCT04488042
Title: Stapler-less Burst Pressure in a Ex-vivo Human Gastric Tissue: a Randomized Controlled Trial
Brief Title: Stapler-less Burst Pressure in a Ex-vivo Human Gastric Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Claudio Gambardella, Researcher, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Stapler-less sleeve
Record Dates: First submitted 2020-07-22; First posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Obesity, Morbid; Suture, Complication; Suture Rupture
Keywords: Sleeve gastrectomy; stapler-less; burst pressure; leaks
MeSH Terms: conditions — Obesity, Morbid | interventions — Sutures

STUDY DESIGN:
Intervention Model Description: the gastric specimen were immediately randomly allocated to the two groups
Who Masked: Participant, Care Provider
Masking Description: Physicians who performed manometry were blinded from specimen allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stapler-less (Experimental): after the LSG stapler line removal by electrothermal bipolar-activated device (LigaSure Atlas™, Valleylab, Boulder, CO, USA), a stapler-less hand-sewn reconstruction was adopted. A single extra-mucosal running barbed suture (3/0 V-Loc™ suture; Covidien, Mansfield, MA, USA), incorporating sero- and submucosal gastric layers, closed the gastric tube.
  Interventions: Other: Stapler-less gastrectomy
- Conventional Stapler (Active Comparator): no reinforcement was performed, the stomach was re-sleeved along a 40F bougie with Echelon Flex Endopath 60-mm linear stapler (Ethicon Endo-Surgery, Cincinnati, OH, USA) to reproduce standard volume of remnant LSG stomach and/or eliminating zig-zag shape of suture-line.
  Interventions: Other: Suture

INTERVENTIONS:
Other: Stapler-less gastrectomy — After the LSG stapler line removal by electrothermal bipolar-activated device (LigaSure Atlas™, Valleylab, Boulder, CO, USA), a stapler-less hand-sewn reconstruction was adopted. A single extra-mucosal running barbed suture (3/0 V-Loc™ suture; Covidien, Mansfield, MA, USA), incorporating sero- and submucosal gastric layers, closed the gastric tube.
  Arms: Stapler-less
Other: Suture — No reinforcement was performed, the stomach was re-sleeved along a 40F bougie with Echelon Flex Endopath 60-mm linear stapler (Ethicon Endo-Surgery, Cincinnati, OH, USA) to reproduce standard volume of remnant LSG stomach and/or eliminating zig-zag shape of suture-line.
  Arms: Conventional Stapler

SUMMARY:
Stapler-less laparoscopic sleeve gastrectomy (LSG) is emerging as a new potential affordable cost-effective alternative procedure. However, no pre-clinical data are currently available on human tissue. We aimed to evaluate whether traditionally suturing without the use of surgical stapling may produces a comparable bursting pressure on human gastric tissue.

DETAILED DESCRIPTION:
Stapler-less laparoscopic sleeve gastrectomy (LSG) is emerging as a new potential affordable cost-effective alternative procedure. However, no pre-clinical data are currently available on human tissue. We aimed to evaluate whether traditionally suturing without the use of surgical stapling may produces a comparable bursting pressure on human gastric tissue.

A prospective cohort of consecutive patients underwent LSG was divided in two groups to compare a barbed extramucosal running suture (stapler-less) versus a standard stapler line. A burst pressure test was applied to the gastric specimen employing high-resolution manometric catheter. Type, location and features of the leak were described.

In human ex-vivo model, traditional surgical suture (i.e. running hand-sewn) produced an effective temporary closure, with superior resistance to increasing volume and pressure. How this may impact on clinical LSG outcomes needs further evaluations and was not the object of this study.

ELIGIBILITY:
Inclusion Criteria:

* Morbid obesity according to IFSO guidelines

Exclusion Criteria:

* Gastric specimen with injury and/or electrocoagulation signs at serosa
* Presence of comorbidities capable of affecting specimen tissue resistance (i.e. type II diabetes, gastric ulcer, connective tissue disease, systemic sclerosis, polymyositis)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Gastric specimen tissue resistance | During procedure
  Evaluate the manometric burst pressure in the ex-vivo gastric specimen after hand-sewn running suture (group 1), and stapler suturing (group 2)
Gastric specimen volume resistance | During procedure
  the saline volume needed to determine a gastric leak in the ex-vivo gastric specimen after hand-sewn running suture (group 1), and stapler suturing (group 2)

CONTACTS AND LOCATIONS:
Overall Officials: Gianmattia del Genio, Prof, Principal Investigator — University of Campania Luigi Vanvitelli
Locations (1):
- Claudio Gambardella, Naples, Italy

IPD SHARING:
Plan to Share IPD: No